CLINICAL TRIAL: NCT02867475
Title: Physical Activity in Patients With Cancer: Epidemiological Study of Patients' Beliefs and Promotional Messages Efficiency
Brief Title: REduction of Physical Inactivity Facing the CAncer
Acronym: RESCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013/03 RESCA; 2013-A01015-40 (Other: ANSM ID RCB)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Physical activity motivation
  Interventions: Other: Physical activity motivation

INTERVENTIONS:
Other: Physical activity motivation — Physical activity motivation

SUMMARY:
Study 1:

The investigator hypothesizes that the level of knowledge about the benefits of physical activity, physical activity level and physical fatigue level observed in cancer patients, would influence their beliefs about physical activity and their intention to engage in AP.

DETAILED DESCRIPTION:
Study 2:

Because of a recent research, it is shown that a narrative message from a peer generates an identification, a sense of self-efficacy and intention to practice in sedentary patients with breast cancer.

The investigator hypothesize that a promotional message about physical activity, issued by a self-determined peer (intrinsic motivation), compared to a non-self-determined peer (extrinsic motivation), generate higher scores of positive beliefs about physical activity and intention to engage in a physical activity program for sedentary patients.

These promotional messages will be delivered through two videos, one featuring the self-determined pair, the other featuring the non-self-determined pair.

ELIGIBILITY:
Inclusion Criteria:

* PS 0-3
* Patients with breast cancer undergoing chemotherapy treatment
* neoadjuvant, adjuvant, metastatic, any histological type, any stage breast cancer
* Sedentary Patients (physical activity score of Dijon less than or equal to 20)

Exclusion Criteria:

* Patients with PS greater than 3
* Patients with cognitive disorders not allowing them to understand the questionnaires and study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
CaBES | 1 day
  psychometric measures: Cancer Beliefs and Exercise Scale Questionnaire

SECONDARY OUTCOMES:
Multidimensional Fatigue Inventory | 1 day
  Fatigue level determination
Dijon's Score | 1 day
  Physical activity level determination

CONTACTS AND LOCATIONS:
Overall Officials: Véronique MARI, md, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine LACASSAGNE, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided